CLINICAL TRIAL: NCT01891006
Title: Intervention for Postpartum Infections Following Caesarean Section - a Randomized Controlled Trial
Brief Title: Intervention for Postpartum Infections Following Caesarean Section
Acronym: APIPICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other); Hvidovre University Hospital (Other); Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Nana Hyldig, PhD Student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20120163
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Surgical Wound Infection; Infection; Cesarean Section; Cesarean Section; Dehiscence; Complications; Cesarean Section; Complications; Cesarean Section, Wound, Dehiscence; Wound; Rupture, Surgery, Cesarean Section
Keywords: Randomized Controlled Trial; Economical Evaluation; Caesarean Section; Cesarean Section; Postoperative Wound Treatment; Surgical Site Infections; Wound Infections; Infectious Morbidity; Negative Pressure Wound Therapy
MeSH Terms: conditions — Surgical Wound Infection; Infections; Wounds and Injuries; Rupture; Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): Negative Pressure Wound Therapy (NPWT) is an alternative method of conservative wound management, which uses negative pressure to promote wound healing in both chronic and acute wounds. The rationale for using NPWT is that it mechanically stimulates the formation of new tissue and removes wound fluid and infectious material
  Interventions: Device: Negative Pressure Wound Therapy
- A standard wound dressing (Other): The standard wound dressing is a hydrofiber or alginate dressing, used for open wound
  Interventions: Other: Standard wound dressing

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — The Negative Pressure Wound Therapy are changed on the 2. day and removed on the 4. day after the re-operation.
  Other Names: RENASYS-G from Smith&Nephew
  Arms: Negative Pressure Wound Therapy
Other: Standard wound dressing — The standard wound dressing is a a hydrofiber or alginate dressing used for open wounds
  Arms: A standard wound dressing

SUMMARY:
The purpose of this study is to examine whether Negative Pressure Wound Therapy is an effective wound treatment compared to conventional wound treatment in the period of time from reoperation to re-suturing in women having surgical wound rupture after Caesarean Section.

DETAILED DESCRIPTION:
This study is a non-blinded randomized controlled trial and a concurrent Health Economic. The study examines the effect on wound healing using NPWT compared with conventional wound treatment in women, who experience spontaneous dehiscence or where a surgeon deliberately opens the wound after Caesarean Section (CS).

Women, who have given informed consent, will be randomized to either intervention or control group via a computer-generated randomization program. It is not possible to blind either participants or therapists. The analysis will be carried out on an intention to treat basis.

Women with post-CS wound infection will be hospitalized and the wound will be reopened and cleaned under general anaesthesia. In the intervention group women will be treated with NPWT. The change of wound dressing on the second day takes place in the obstetrical or plastic surgery ward. On the fourth day, the NPWT material will be removed and the wound evaluated before re-suturing. In the control group the wound will be treated with a hydrofiber or alginate dressing. Changes of wound dressing will take place on the second and fourth days as in the intervention group. In both groups, when the wound is evaluated on the second and fourth day, it will be described and measured (depth, width, length). After four days of treatment, the wound will be re-sutured in both groups. It is expected that some wounds are not suitable for re-suturing on the fourth day. If a woman does not want to participate, she will receive the conventional treatment, which corresponds to the treatment in the control group. Women, who do not wish to participate, will be asked for permission to use their data in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Women, who can read and understand Danish

Exclusion Criteria:

* Serious illness requiring medical treatment, such as cancer
* Stillborn child
* If the fascia is ruptured

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The frequency of re-rupture in each study group | Within the first 30 days after surgery

SECONDARY OUTCOMES:
Length of hospitalization | Within the first 30 days after Caesarean Section
Readmission to hospital due to wound complications after the re-operation | Within the first 30 days after Caesarean Section
Number of participants with a decreased health-related quality of life score as a measure of satisfaction and tolerability | Within the first 30 days after Caesarean Section
  A health-related quality of life measure, recorded in Quality Adjusted Life Years at the two interventions. The health-related quality of life score is measured on the 4 day after the re-operation and at the 6 and 12 months follow-up.
The cosmetic outcome as a measure of satisfaction | A 6 and 12 months follow-up
  The scar will be evaluated by a plastic surgeon at a clinical examination 6 and 12 months after the re-operation. After study completion pictures of the scars will be evaluated by two blinded plastic surgeons, using two predefined scar scales.

CONTACTS AND LOCATIONS:
Overall Officials: Nana Hyldig, PhD Student, Study Chair — Odense University Hospital, department of Plastic Surgery, University of Southern Denmark, Faculty of Health Sciences, institute of Clinical Research, research unit, department of Gynaecology and Obstetrics
Locations (1):
- Odense University Hospital, Odense, Denmark